CLINICAL TRIAL: NCT04593004
Title: Randomized Open-Label Trial Comparing Teledermatology vs. Face-to-Face Consultation in the Follow-Up of Patients With Mild-to-Moderate Acne
Brief Title: Teledermatology vs. Face-to-Face Visits in the Follow-Up of Patients With Acne
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2019-00620
Record Dates: First submitted 2020-10-09; First posted 2020-10-19 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Acne Vulgaris
Keywords: acne; telemedicine; teledermatology
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Intervention Model Description: 1:1 stratified random allocation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Teledermatology (Experimental)
  Interventions: Device: Teledermatology
- Face-to-face consultation (Active Comparator)
  Interventions: Other: Face-to-face consultation

INTERVENTIONS:
Device: Teledermatology — Patients will be assessed and followed-up by trained physicians through a store-and-forward system (teledermatology online service - Evita® app), which allows patients to upload pictures of skin areas affected by acne as well as their symptoms or questions related to their disease.
  Arms: Teledermatology
Other: Face-to-face consultation — Patients will be assessed and followed-up by trained physicians through regular face-to-face outpatient consultations.
  Arms: Face-to-face consultation

SUMMARY:
Acne vulgaris is a common cutaneous inflammatory condition of sebaceous follicles that can profoundly affect patients' quality of life, especially at a young age. In this context the use of teledermatology can potentially reduce the healthcare costs associated to traditional consultations as well as the costs related to travel and loss of school/working time for the patient, with a clear benefit for the whole community. Since 2016, the Department of Dermatology at Inselspital Hospital in Bern has a portal and a smartphone app for online advice service.

Hereby the investigators propose to explicitly investigate the efficacy of this system in reducing healthcare costs as compared to traditional face-to-face consultations, in a cohort of patients with mild-to-moderate acne vulgaris.

ELIGIBILITY:
Inclusion Criteria:

* Given written informed consent
* Mild-to-moderate acne as assessed by IGA scale
* Willingness and ability to adhere the study protocol

Exclusion Criteria:

* Need for systemic therapy for acne with Isotretinoin
* Inability to use the teledermatology system

Ages: 18 Years to 28 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2020-10-07 (Actual); Primary Completion 2022-06-20 (Actual); Study Completion 2022-06-20 (Actual)

PRIMARY OUTCOMES:
Total time spent by dermatologist after baseline | 4 months
  Total cumulative time spent by dermatologist for face-to-face consultations or online assessments after baseline.

SECONDARY OUTCOMES:
Total time spent by patient after baseline | 4 months
  Total cumulative time spent by patient for visit-related travels and/or online procedures after baseline.
Acne severity improvement | 2, 4 and 6 months
  Acne severity improvement from baseline as assessed by 5-point ordinal investigator's global assessment (IGA) scale, ranging from 1 to 5, with higher scores indicating a worse outcome.
Number of therapies prescribed for acne | 2, 4 and 6 months
Patient study satisfaction | 6 months
  Overall patient satisfaction regarding the service received during the study as assessed by 11-point anchored visual analogue scale (VAS), ranging from 0 to 10, with higher scores indicating a better outcome.
Patient quality of life improvement | 6 months
  Patient quality of life improvement from baseline as assessed by dermatology life quality index (DLQI), ranging from 0 to 30, with higher scores indicating a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Hunger, MD, Principal Investigator — Insel Gruppe AG, University Hospital Bern
Locations (1):
- Department of dermatology, University Hospital Inselspital, Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No